CLINICAL TRIAL: NCT00761904
Title: A Study Assessing the Effect of Cardiovascular Medications Provided as Low-cost, Evidence-based Generic Samples
Brief Title: The Effect of Providing Free Samples of Generic Cardiovascular Medications to Physicians
Acronym: SAMPLES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: William H. Shrank MD MSHS, Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 08-001010; 1K23HL090505-01 (NIH)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Hypertension; Hyperlipidemia
Keywords: hypertension; hyperlipidemia; free generic samples
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Hydrochlorothiazide; Simvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- receipt of free generic samples (Experimental)
  Interventions: Behavioral: Free Generic Samples (hydrochlorothiazide, simvastatin)
- usual prescribing (No Intervention)

INTERVENTIONS:
Behavioral: Free Generic Samples (hydrochlorothiazide, simvastatin) — Free samples of generic hydrochlorothiazide (12.5 mg tabs) and simvastatin (20 mg tabs)
  Arms: receipt of free generic samples

SUMMARY:
In this randomized controlled trial, we will provide primary care physicians with free samples of highly effective generic cardiovascular medications. We will test whether this intervention will stimulate cost-effective prescribing, reducing drug costs and improving adherence to essential cardiovascular medications.

DETAILED DESCRIPTION:
Highly-effective generic cardiovascular medications are frequently underused, leading to greater overall drug costs and cost-related non-adherence. Interventions are needed to stimulate appropriate generic drug use without creating administrative or financial barriers to branded medications that may impede essential medication use.

The SAMPLES trial is a clustered, randomized controlled trial of the effect of providing physicians with free generic samples of hydrochlorothiazide for hypertensive patients and simvastatin for patients with hyperlipidemia. We will randomize 660 primary care physicians in Pennsylvania, clustered by physician practice, to receive free samples for both conditions or to receive no samples. We will use pharmacy claims of their patient population enrolled in a state-sponsored prescription drug assistance program to evaluate outcomes of interest. The primary outcomes are physician prescribing behavior (proportion of prescriptions that are generic), and patient adherence to chronic therapy. Secondary outcomes will include physician adherence to established guidelines (for anti-hypertensive regimens) and overall prescription drug costs. Primary analyses will be based on intention-to-treat principles.

This trial highlights a new and innovative approach to stimulate cost-effective prescribing. Free generic samples can reduce overall drug costs as well as out-of-pocket costs to the patient without sacrificing efficacy, and may result in improved adherence to essential cardiovascular medications. This intervention may also improve adherence to practice guidelines and improve the quality of care received. If found to be effective, this strategy could be utilized broadly by private insurers or government payers aiming to stimulate more cost-effective and higher-quality care.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians receiving an existing academic detailing program in Pennsylvania

Exclusion Criteria:

* Those with administrative policies stating they do not accept free samples

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of prescriptions filled for generic medications | 6 months after receipt of samples
Patient adherence - Amount of prescriptions actually filled (Proportion of Days Covered) within each class in the first year of use of an anti-hypertensive or lipid-lowering medication | in the year subsequent to patient initiation of an anti-hypertensive or lipid-lowering medication

SECONDARY OUTCOMES:
The sum of medication costs for all prescriptions used to treat either hypertension or hypercholesterolemia. | The year before and the year after provision of samples
Guideline adherence - Proportion of patients who received first-line anti-hypertensive medications suggested by JNC-VII when medications are initiated. | In the 6 months after receipt of samples

CONTACTS AND LOCATIONS:
Overall Officials: William H Shrank, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States